CLINICAL TRIAL: NCT02969863
Title: The Monitoring Study: Evaluating the Effect of Remote Monitoring For Hypoglycemia on Bionic Pancreas Safety and Efficacy
Brief Title: The Monitoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002450
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Type1diabetes
Keywords: bionic pancreas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Usual Care Arm - Monitored (Active Comparator): Subjects will manage their own diabetes and will wear a blinded Dexcom G4 CGM to record their glucose data during the week. They will be monitored for CGM connectivity and hypoglycemia.
  Monitored for hypoglycemia
  Interventions: Other: Monitored for Hypoglycemia
- Usual Care Arm - Unmonitored (Active Comparator): Subjects will manage their own diabetes and will wear a blinded Dexcom G4 CGM to record their glucose data during the week. They will be monitored only for CGM connectivity, not hypoglycemia.
  Not monitored for hypoglycemia
  Interventions: Other: Not Monitored for Hypoglycemia
- Bihormonal Bionic Pancreas - Monitored (Experimental): Subjects will wear the bihormonal bionic pancreas, consisting of a Dexcom G4 CGM, an insulin and glucagon pump and an iPhone running the study algorithm. They will be monitored for CGM connectivity and hypoglycemia.
  Monitored for hypoglycemia
  Interventions: Device: Bihormonal Bionic Pancreas; Other: Monitored for Hypoglycemia
- Bihormonal Bionic Pancreas - Unmonitored (Experimental): Subjects will wear the bihormonal bionic pancreas, consisting of a Dexcom G4 CGM, an insulin and glucagon pump and an iPhone running the study algorithm. They will be monitored only for CGM connectivity, not hypoglycemia.
  Not monitored for hypoglycemia
  Interventions: Device: Bihormonal Bionic Pancreas; Other: Not Monitored for Hypoglycemia
- Insulin Only Bionic Pancreas - Monitored (Experimental): Subjects will wear the insulin only bionic pancreas, consisting of a Dexcom G4 CGM, an insulin pump, and an iPhone running the study algorithm. They will be monitored for CGM connectivity and hypoglycemia.
  Monitored for hypoglycemia
  Interventions: Device: Insulin Only Bionic Pancreas; Other: Monitored for Hypoglycemia
- Insulin Only Bionic Pancreas - Unmonitored (Experimental): Subjects will wear the insulin only bionic pancreas, consisting of a Dexcom G4 CGM, an insulin pump, and an iPhone running the study algorithm. They will be monitored only for CGM connectivity, not hypoglycemia.
  Not monitored for hypoglycemia
  Interventions: Device: Insulin Only Bionic Pancreas; Other: Not Monitored for Hypoglycemia

INTERVENTIONS:
Device: Bihormonal Bionic Pancreas — Participants will wear a Bionic Pancreas that uses glucagon and insulin (bihormonal) to automate their glucose control based on continuous glucose monitor readings.
  Arms: Bihormonal Bionic Pancreas - Monitored; Bihormonal Bionic Pancreas - Unmonitored
Device: Insulin Only Bionic Pancreas — Participants will wear a Bionic Pancreas that uses just insulin (insulin-only) to automate their glucose control based on continuous glucose monitor readings.
  Arms: Insulin Only Bionic Pancreas - Monitored; Insulin Only Bionic Pancreas - Unmonitored
Other: Monitored for Hypoglycemia — During half of the study arms (one each bihormonal bionic pancreas, insulin-only bionic pancreas and usual care) the subjects will be remotely monitored for device connectivity and hypoglycemia, and will be notified by study staff any time their continuous glucose monitor reads less than 50 mg/dl for 15 mintues.
  Arms: Bihormonal Bionic Pancreas - Monitored; Insulin Only Bionic Pancreas - Monitored; Usual Care Arm - Monitored
Other: Not Monitored for Hypoglycemia — During half of the study arms (one each bihormonal bionic pancreas, insulin-only bionic pancreas and usual care) the subjects will be remotely monitored for device connectivity only, not hypoglycemia.
  Arms: Bihormonal Bionic Pancreas - Unmonitored; Insulin Only Bionic Pancreas - Unmonitored; Usual Care Arm - Unmonitored

SUMMARY:
To conduct an outpatient study testing two configurations of the bionic pancreas (bi-hormonal and insulin-only) with and without remote monitoring of hypoglycemia in 25 adult (≥ 18 years of age) subjects with type 1 diabetes in a random-order crossover study versus usual care with an insulin pump with and without remote monitoring of hypoglycemia.

DETAILED DESCRIPTION:
The rationale for this study is to measure the safety of eliminating the glycemic monitoring that the investigators have done in all of the previous outpatient studies under both insulin only and bihormonal bionic pancreas control. The investigators are planning to transition the outpatient studies to an integrated bionic pancreas, the iLet, in the near future. The intended use of this device does not include remote monitoring, which would not be feasible on a commercial scale. Therefore, in this trial the investigators will test the effects on hypoglycemia of eliminating blood glucose related monitoring. In addition, the investigators will perform a pilot trial testing the effects of the bionic pancreas on food intake, exercise, weight and body composition. The primary purpose of this pilot is to assess the feasibility of performing these measurements in the context of a larger trial and to collect data that can be used to power sub-studies of pivotal trials looking at these outcomes. Finally, the investigators will test the accuracy of two new CGM devices to see if they have sufficient accuracy to provide glucose data to the bionic pancreas. If so, this would provide new options for users who may have difficulties with the only currently validated CGM for this purpose, the Dexcom G4 AP / G5 platform.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and have had clinical type 1 diabetes for at least one year managed using an insulin pump for ≥ 6 months
* Prescription medication regimen stable for > 1 month (except for medications that will not affect the safety of the study and are not expected to affect any outcome of the study, in the judgment of the principal investigator)
* Live within a 60 minute drive-time radius of the central monitoring location
* Willing to remain within a 120 minute drive-time radius of the central monitoring location throughout the study
* Have someone over 18 years of age who lives with them, has access to where they sleep, is willing to be in the house when the subject is sleeping, and is willing to receive calls from the study staff and check the welfare of the study subject if telemetry shows a technical problem or severe biochemical hypoglycemia without subject response and the subject does not answer their telephone (up to two individuals can share this role, but they must be willing to carefully coordinate with each other and the subject so that one of them is clearly designated as having this responsibility at any given time)
* Willing to wear one or two infusion sets and one Dexcom CGM sensor and change sets frequently (at least one new glucagon infusion set daily during bi-hormonal arms, and insulin infusion set every other day throughout the study)
* Willing to wear two additional CGM sensors that must be placed in the upper arm

Exclusion Criteria:

* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory, unable to speak and read English)
* Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the subject
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception Subjects must use acceptable contraception for the two weeks prior to the study, throughout the study and for the two weeks following the study.

Acceptable contraception methods include: Oral contraceptive pill (OCP), Intrauterine Device (IUD, hormonal or copper), Male condoms, Female condoms, Diaphragm or cervical cap with spermicide, Contraceptive patch (such as OrthoEvra), Contraceptive implant (such as Implanon, Nexplanon), Vaginal ring (such as NuvaRing), Progestin shot (such as Depo-Provera), Male partner with a vasectomy proven to be effective by semen analysis

* Need to go outside of the designated geographic boundaries during the study
* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days), use of marijuana within 1 month of enrollment, or other substance abuse (use within the last 6 months of controlled substances other than marijuana without a prescription)
* Unwilling or unable to refrain from drinking more than 2 drinks in an hour or more than 4 drinks in a day or use of marijuana during the trial
* Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of beta blockers will be allowed as long as the dose is stable and the subject does not meet the criteria for hypoglycemia unawareness while taking that stable dose, but use of benzodiazepines or narcotics, even if by prescription, may be excluded according to the judgment of the principal investigator)
* History of liver disease that is expected to interfere with the anti-hypoglycemia action of glucagon (e.g. liver failure or cirrhosis). Other liver disease (i.e. active hepatitis, steatosis, active biliary disease, any tumor of the liver, hemochromatosis, glycogen storage disease) may exclude the subject if it causes significant compromise to liver function or may do so in an unpredictable fashion.
* Renal failure on dialysis
* Personal history of cystic fibrosis, pancreatitis, pancreatic tumor, or any other pancreatic disease
* Any known history of coronary artery disease including, but not limited to, history of myocardial infarction, stress test showing ischemia, history of angina, or history of intervention such as coronary artery bypass grafting, percutaneous coronary intervention, or enzymatic lysis of a presumed coronary occlusion)
* Abnormal EKG consistent with coronary artery disease or increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, prior myocardial infarction, proximal LAD critical stenosis (Wellen's sign), prolonged QT interval (> 440 ms). Non-specific ST segment and T wave changes are not grounds for exclusion in the absence of symptoms or history of heart disease. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.
* Congestive heart failure (established history of CHF, lower extremity edema, paroxysmal nocturnal dyspnea, or orthopnea)
* History of TIA or stroke
* Seizure disorder, history of any non-hypoglycemic seizure within the last two years, or ongoing treatment with anticonvulsants
* History of hypoglycemic seizures (grand-mal) or coma in the last year
* History of pheochromocytoma: fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor:

  * Episodic or treatment refractory (requiring 4 or more medications to achieve normotension) hypertension
  * Paroxysms of tachycardia, pallor, or headache
  * Personal or family history of MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease
* History of adrenal disease or tumor
* Hypertension with systolic BP ≥160 mm Hg or diastolic BP ≥100 despite treatment
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
* The presence of any other active implanted device
* Unable to completely avoid acetaminophen for duration of study
* Unable to completely avoid ascorbic acid (Vitamin C) for duration of study
* Unable to completely avoid salicylic acid (used in some pain relievers such as Aspirin and some skin care products)
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study
* History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
* History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
* Use of oral (e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, DPP-4 inhibitors, SGLT-2 inhibitors) anti-diabetic medications
* Lives in or frequents areas with poor Verizon wireless network coverage (which would prevent remote monitoring)
* Any factors that, in the opinion of the principal investigator would interfere with the safe completion of the study
* A condition preventing or complicating the placement, operation or removal of the Senseonics sensor or wearing of transmitter, including upper extremity deformities or skin condition
* Currently receiving (or likely to need during the study period): immunosuppressant therapy, chemotherapy, anticoagulant/antithrombotic therapy (excluding aspirin), glucocorticoids (excluding ophthalmic or nasal). This does include the use of inhaled and topical glucocorticoids and antibiotics for chronic infection
* A condition requiring or likely requiring magnetic resonance imaging (MRI), Computed Tomography (CT) scan, or high-frequency electrical heat (diathermy)
* A known topical or local anesthetic allergy
* A known glucocorticoids allergy
* The presence of any other CGM sensor or transmitter located in the upper arm (other location is acceptable)
* Hemoglobin < 12 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Diabetes Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 subjects were enrolled, but only 24 participated in the study. 2 subjects were ineligible, and 1 could not participate for scheduling reasons. 1 of the 24 was terminated by the investigator during the first arm of the study, so that 1 subject only started 1 arm. 23 subjects finished that arm, and 23 subjects started and finished the other arms
Groups:
- BBPM First, Then BBP, Then UCM, Then UC, Then IOBPM, Then IOBP; UCM First, Then UC, Then IOBPM, Then IOBP, Then BBPM, Then BBP; IOBPM First, Then IOBP, Then BBPM, Then BBP, Then UCM, Then UC; UC First, Then UCM, Then BBP, Then BBPM, Then IOBP, Then IOBPM; IOBP First, Then IOBPM, Then UC, Then UCM, Then BBP, Then BBPM; BBP First, Then BBPM, Then IOBP, Then IOBPM, Then UC, Then UCM: UC=usual care-Subjects will manage their own diabetes and wear a Dexcom CGM G5 to record their glucose data during the week
  IOBP-insulin only bionic pancreas. Subjects will wear the insulin only bionic pancreas consisting of a Dexcom G5 CGM, an insulin pump, and an iPhone running the study algorithm.
  BBP- bihormonal bionic pancreas- Subjects will wear the bihormonal bionic pancreas, consisting of a Dexcom G5 CGM, and insulin and glucagon pump and an iPhone running the study algorithm
  M-arm includes real-time remote monitoring for hypoglycemia
Period: Overall Study
Arm/Group | BBPM First, Then BBP, Then UCM, Then UC, Then IOBPM, Then IOBP | UCM First, Then UC, Then IOBPM, Then IOBP, Then BBPM, Then BBP | IOBPM First, Then IOBP, Then BBPM, Then BBP, Then UCM, Then UC | UC First, Then UCM, Then BBP, Then BBPM, Then IOBP, Then IOBPM | IOBP First, Then IOBPM, Then UC, Then UCM, Then BBP, Then BBPM | BBP First, Then BBPM, Then IOBP, Then IOBPM, Then UC, Then UCM
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4 | 4 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who began participating in the study
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Hemoglobin A1c [Mean (Standard Deviation); unit: percent] | 7.2 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent With Dexcom CGMG < 60 mg/dl
Description: A measure of hypoglycemia capturing amount of time the continuous glucose monitor is reading less than 60 mg/dl
Time Frame: days 2-7
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Usual Care Arm - Monitored: Subjects will manage their own diabetes and will wear a blinded Dexcom G4 CGM to record their glucose data during the week. They will be monitored for CGM connectivity and hypoglycemia.
  Monitored for hypoglycemia
  Monitored for Hypoglycemia: During half of the study arms (one each bihormonal bionic pancreas, insulin-only bionic pancreas and usual care) the subjects will be remotely monitored for device connectivity and hypoglycemia, and will be notified by study staff any time their continuous glucose monitor reads less than 50 mg/dl for 15 mintues.
- Usual Care Arm - Unmonitored: Subjects will manage their own diabetes and will wear a blinded Dexcom G4 CGM to record their glucose data during the week. They will be monitored only for CGM connectivity, not hypoglycemia.
  Not monitored for hypoglycemia
  Not Monitored for Hypoglycemia: During half of the study arms (one each bihormonal bionic pancreas, insulin-only bionic pancreas and usual care) the subjects will be remotely monitored for device connectivity only, not hypoglycemia.
- Bihormonal Bionic Pancreas - Monitored: Subjects will wear the bihormonal bionic pancreas, consisting of a Dexcom G4 CGM, an insulin and glucagon pump and an iPhone running the study algorithm. They will be monitored for CGM connectivity and hypoglycemia.
  Monitored for hypoglycemia
  Bihormonal Bionic Pancreas: Participants will wear a Bionic Pancreas that uses glucagon and insulin (bihormonal) to automate their glucose control based on continuous glucose monitor readings.
  Monitored for Hypoglycemia: During half of the study arms (one each bihormonal bionic pancreas, insulin-only bionic pancreas and usual care) the subjects will be remotely monitored for device connectivity and hypoglycemia, and will be notified by study staff any time their continuous glucose monitor reads less than 50 mg/dl for 15 mintues.
- Bihormonal Bionic Pancreas - Unmonitored: Subjects will wear the bihormonal bionic pancreas, consisting of a Dexcom G4 CGM, an insulin and glucagon pump and an iPhone running the study algorithm. They will be monitored only for CGM connectivity, not hypoglycemia.
  Not monitored for hypoglycemia
  Bihormonal Bionic Pancreas: Participants will wear a Bionic Pancreas that uses glucagon and insulin (bihormonal) to automate their glucose control based on continuous glucose monitor readings.
  Not Monitored for Hypoglycemia: During half of the study arms (one each bihormonal bionic pancreas, insulin-only bionic pancreas and usual care) the subjects will be remotely monitored for device connectivity only, not hypoglycemia.
- Insulin Only Bionic Pancreas - Monitored: Subjects will wear the insulin only bionic pancreas, consisting of a Dexcom G4 CGM, an insulin pump, and an iPhone running the study algorithm. They will be monitored for CGM connectivity and hypoglycemia.
  Monitored for hypoglycemia
  Insulin Only Bionic Pancreas: Participants will wear a Bionic Pancreas that uses just insulin (insulin-only) to automate their glucose control based on continuous glucose monitor readings.
  Monitored for Hypoglycemia: During half of the study arms (one each bihormonal bionic pancreas, insulin-only bionic pancreas and usual care) the subjects will be remotely monitored for device connectivity and hypoglycemia, and will be notified by study staff any time their continuous glucose monitor reads less than 50 mg/dl for 15 mintues.
- Insulin Only Bionic Pancreas - Unmonitored: Subjects will wear the insulin only bionic pancreas, consisting of a Dexcom G4 CGM, an insulin pump, and an iPhone running the study algorithm. They will be monitored only for CGM connectivity, not hypoglycemia.
  Not monitored for hypoglycemia
  Insulin Only Bionic Pancreas: Participants will wear a Bionic Pancreas that uses just insulin (insulin-only) to automate their glucose control based on continuous glucose monitor readings.
  Not Monitored for Hypoglycemia: During half of the study arms (one each bihormonal bionic pancreas, insulin-only bionic pancreas and usual care) the subjects will be remotely monitored for device connectivity only, not hypoglycemia.
Arm/Group | Usual Care Arm - Monitored | Usual Care Arm - Unmonitored | Bihormonal Bionic Pancreas - Monitored | Bihormonal Bionic Pancreas - Unmonitored | Insulin Only Bionic Pancreas - Monitored | Insulin Only Bionic Pancreas - Unmonitored
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23
percentage of time | 1.32 (1.39) | 1.95 (2.11) | 1.05 (1.01) | 0.99 (0.93) | 1.55 (1.16) | 1.66 (1.33)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Usual Care Arm - Monitored | Usual Care Arm - Unmonitored | Bihormonal Bionic Pancreas - Monitored | Bihormonal Bionic Pancreas - Unmonitored | Insulin Only Bionic Pancreas - Monitored | Insulin Only Bionic Pancreas - Unmonitored
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Arm - Monitored (N=24) | Usual Care Arm - Unmonitored (N=24) | Bihormonal Bionic Pancreas - Monitored (N=24) | Bihormonal Bionic Pancreas - Unmonitored (N=24) | Insulin Only Bionic Pancreas - Monitored (N=24) | Insulin Only Bionic Pancreas - Unmonitored (N=24)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The subject reported a hypoglycemic event that he was not called for. Remote monitoring did not see this or notify study staff. The subject reported that he treated using oral carbohydrates, and it resolved without incident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT02969863/Prot_SAP_000.pdf